CLINICAL TRIAL: NCT00792246
Title: Define the Pharmacokinetics of Oral Voriconazole in Children With Extensive Gastrointestinal Graft Versus Host Disease
Brief Title: Voriconazole Pharmacokinetics in Children With Gastrointestinal Graft Versus Host Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phillip Brian Smith (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Phillip Brian Smith, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00004318
Record Dates: First submitted 2008-11-13; First posted 2008-11-17 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Graft Versus Host Disease; Stem Cell Transplantation
Keywords: pharmacokinetics; pediatric; bioavailability
MeSH Terms: conditions — Graft vs Host Disease | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- graft versus host disease (Experimental): Patients receiving oral voriconazole will be switched to intravenous voriconazole. Pharmacokinetics will be determined after each formulation.
  Interventions: Drug: voriconazole
- No graft versus host disease (Experimental): Patients receiving oral voriconazole will be switched to intravenous voriconazole. Pharmacokinetics will be determined after each formulation.
  Interventions: Drug: voriconazole

INTERVENTIONS:
Drug: voriconazole — Voriconazole formulation will be changed from oral to intravenous at the same dose the subject is currently receiving per standard of care.
  Arms: graft versus host disease
Drug: voriconazole — Voriconazole formulation will be changed from oral to intravenous at the same dose the subject is currently receiving per standard of care.
  Arms: No graft versus host disease

SUMMARY:
Determine how much voriconazole is absorbed when the product is given by mouth to children with extensive graft versus host disease after a stem cell transplantation and determine the correct dosing of voriconazole in this population.

Hypothesis: Children with gastrointestinal graft versus host disease will have decreased absorption of oral voriconazole and require higher doses of voriconazole in order to prevent or treat fungal infections.

DETAILED DESCRIPTION:
Disseminated fungal infections are a leading cause of mortality in children who receive hematopoietic stem cell transplantation (SCT). Therefore, children routinely receive prophylactic and empirical antifungal therapy after SCT. The most commonly used antifungal agent in this population is voriconazole. Voriconazole can be given via intravenous or oral routes and children who are post SCT are routinely switched from the intravenous to oral formulation at the time of hospital discharge. However, the absorption and systemic exposure of oral voriconazole has not been well-described in children. Furthermore, many children who undergo transplantation develop gastrointestinal graft versus host disease and this likely impacts oral absorption. The magnitude of effect resulting from graft versus host disease on absorption of voriconazole and subsequent blood concentrations in children is unknown. Thus children with graft versus host disease are at a particularly high risk of inadequate absorption with subsequent sub-therapeutic levels of voriconazole. They may need higher or more frequent dosing to achieve therapeutic levels. The purpose of my research project is to define the pharmacokinetics of oral voriconazole and establish dosing guidelines in children following SCT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 18 years, sufficient venous access to permit administration of voriconazole, ability to take oral medications, written informed consent provided by the parent or legally authorized representative, and Grade II or higher (extensive) gastrointestinal graft versus host disease for those patients in the graft versus host disease patient subset.

Exclusion Criteria:

* History of anaphylaxis attributed to voriconazole or other triazole compounds, any concomitant condition, which in the opinion of the investigator would preclude a patient's participation in the study, or previous participation in this study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2008-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Reduced bioavailability of oral voriconazole in pediatric patients status post stem cell transplantation with gastrointestinal graft versus host disease | one year

SECONDARY OUTCOMES:
Pharmacokinetics(including clearance, maximum concentration, area under the time concentration curve, and half life) of voriconazole in pediatric patients status post hematopoietic stem cell transplantation. | one year

CONTACTS AND LOCATIONS:
Overall Officials: P Brian Smith, MD, Principal Investigator — Duke Unviersity Medical Center
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States